CLINICAL TRIAL: NCT03631693
Title: The Use of Non-invasive Thermal and Geometrical Surface Imaging on Postoperative Healing Patterns Following Routine Surgical Procedures Used for the Treatment of Periodontal Disease
Brief Title: Imaging Analysis Following Periodontal Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17/LO/1428
Record Dates: First submitted 2018-06-07; First posted 2018-08-15 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Healing Wound; Periodontitis
Keywords: postoperative healing
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Single centre, randomised, single-blind, parallel-group clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The calibrated examiners will be blinded to the study treatment. Samples will be labelled anonymously with subject ID and without codes relating to treatment group; therefore, all sample analyses will be blinded.
  Blinding of the statistician will also take place. Data will be coded during data entry according to treatment group with a number disallowing group identification during analyses. Code details of which each treatment group will be revealed only once analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified papilla preservation flap (Active Comparator): PERIODONTAL SURGICAL INTERVENTION:The first arm is the simplified papilla preservation flap (SPPF) surgery.At visit 3, the SPPF surgery is performed. 2D and 3D imaging on surgical site will be carried out pre and post surgery. 2D and 3D imaging performed on surgical site for all post operative visits.
  Interventions: Procedure: Simplified papilla preservation flap
- Resective flap with osseous recontouring (Active Comparator): PERIODONTAL SURGICAL INTERVENTION: The second arm is the Resective periodontal flap with osseous recontouring (RPFO). At visit 3, the RPFO surgery is performed. 2D and 3D imaging on surgical site will be carried out pre and post surgery. 2D and 3D imaging performed on surgical site for all post operative visits.
  Interventions: Procedure: Resective periodontal flap with osseous recontouring

INTERVENTIONS:
Procedure: Simplified papilla preservation flap — The simplified papilla preservation flap (SPPF) surgery is a conservative surgical procedure aimed at the preservation of the tissues between the teeth providing access for the debridement of the root surface in sites with residual pockets.
  Other Names: SPPF
  Arms: Simplified papilla preservation flap
Procedure: Resective periodontal flap with osseous recontouring — The Resective periodontal flap with osseous recontouring (RPFO) is a surgical procedure that achieves predictable pocket depth reduction by soft and hard tissue resection to obtain a more convenient soft and hard tissue architecture for oral hygiene.
  Other Names: RPFO
  Arms: Resective flap with osseous recontouring

SUMMARY:
This is a single centre, randomised, single-blind, parallel-group clinical trial that aims at evaluating the use of imaging (2D and 3D) in obtaining geometric and thermometric changes of postoperative healing patterns and comorbidities (facial swelling, oedema and inflammation) following two routine surgical procedures performed for the treatment of periodontal (gum) disease.

DETAILED DESCRIPTION:
A surgery in a posterior sextant will be performed per patient. The surgical procedures being compared for their post-operative healing patterns are:

1. Simplified Papilla Preservation Flap (SPPF) which is a conservative flap aiming at preserving the tissues between teeth.
2. Resective Periodontal Flap with Osseous Recontouring (RPFO) which is a conventional surgery which involves hard and soft tissues resection.

Geometric (3D) surface imaging and thermal (2D) surface imaging will be used to assess the post-operative healing patterns and comorbidities (facial swelling, oedema and inflammation) following either of the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy males and females ≥ 30 years of age.
2. Participants must be willing to read, and sign a copy of the "Informed Consent Form" (ICF) form after reading the, "Patient Information Leaflet" (PIS), and after the nature of the study has been fully explained.
3. Participants must present with clinical and radiographic evidence of periodontitis, with one interdental area of Periodontal Pocket Depth (PPD) ≥6mm, Bleeding On Probing (BOP), and Clinical Attachment Level (CAL) ≥6mm in any posterior sextant of their mouth (excluding third molars and the distal aspect of the second molars), or multiple sites (≥9) with PPD ≥5mm, BOP, and CAL ≥5mm.
4. Participants must have completed a course of non-surgical periodontal therapy within 2 years prior to study commencement and have had maintenance including subgingival debridement within 6 months prior to assessment for eligibility.

Exclusion Criteria:

1. Medical history including diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases e.g. cardiovascular disease or AIDS.
2. Antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam.
3. History of alcohol or drug abuse.
4. Self-reported pregnancy or lactation.
5. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration that may interfere with the interpretation of the data.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Geometrical (3D) imaging in post-periodontal surgery wound healing. | Period from pre-surgery to 90 days post-surgery
  Subtracted images from the baseline will identify the area and magnitude of the swelling (changes in volume) in the area of surgery (extra and intra orally).
Thermal (2D) imaging in post-periodontal surgery wound healing. | Period from pre-surgery to 90 days post-surgery
  Subtracted thermography images from the baseline will identify the change of the tissue temperature in the area of surgery (extra and intra orally).

SECONDARY OUTCOMES:
Patient related outcome measures (PROMs) particularly on oral health related quality of life | Period from pre-surgery to 90 days post-surgery
  The secondary objective of this study is to evaluate the impact of the two surgical procedures on patient related outcome measures (PROMs). The Oral impact on daily performances index (OIDP) is going to be used to evaluate health and treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Donos, Prof., Study Director — Institute of Dentistry, QMUL; Nikos Donos, Prof., Principal Investigator — Institute of Dentistry, QMUL
Locations (1):
- Queen Mary University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No